CLINICAL TRIAL: NCT05601219
Title: A Phase 1, Open-Label, Multicenter Study of ADA-011 as Monotherapy and in Combination With a Checkpoint Inhibitor for Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ADA-011 for Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal company decision (non-safety related)
Sponsor: Adanate, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADA-011-001
Record Dates: First submitted 2022-10-17; First posted 2022-11-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: Non-randomized dose escalation followed by dose expansion.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADA-011 Monotherapy Dose Escalation (Experimental): ADA-011 monotherapy will be administered intravenously (IV), every 3 weeks (Q3W) at escalating doses starting with Cycle 1, Day 1, until participant withdrawal. Participants enroll with histologically or cytologically confirmed solid tumors.
  Interventions: Drug: ADA-011
- ADA-011 Monotherapy Dose Expansion (Experimental): ADA-011 monotherapy with the preliminary recommended phase 2 dose (RP2D) of ADA-011, in participants with histologically or cytologically confirmed solid tumors.
  Interventions: Drug: ADA-011
- Combination Therapy Dose Escalation (Experimental): Combination therapy with ADA-011 and PD(L)-1 inhibitor (at escalating ADA-011 doses) will be administered IV Q3W, starting with Cycle 1, Day 1 in participants with histologically or cytologically confirmed solid tumors.
  Interventions: Drug: ADA-011; Drug: PD(L)-1 inhibitor

INTERVENTIONS:
Drug: ADA-011 — ADA-011 will be administered intravenously (IV) Q3W on a 21-day cycle.
Drug: PD(L)-1 inhibitor — PD(L)-1 inhibitor will be administered intravenously (IV) Q3W.
  Arms: Combination Therapy Dose Escalation

SUMMARY:
This study consists of dose escalation evaluation to determine the safety and tolerability of ADA-011 as a monotherapy. Following dose escalation, one or more dose expansion cohorts in selected indications will be explored to further evaluate the safety, tolerability, and preliminary efficacy of ADA-011.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable or metastatic solid tumor that is advanced (nonresectable) or recurrent and progressing since the last antitumor therapy and for which no recognized standard therapy exists
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Measurable disease per RECIST v1.1 or per other criteria best suited for the specific tumor type being evaluated
* Adequate organ function

Exclusion Criteria:

* Treatment with any local or systemic antineoplastic therapy (including chemotherapy, hormonal therapy, or radiation) within 2 weeks prior to the first dose of ADA-011
* Chronic use of corticosteroids in excess of 10 mg daily of prednisone or equivalent within 4 weeks prior to the first dose of ADA-011
* Major trauma or major surgery within 4 weeks prior to the first dose of ADA-011
* AEs from prior anticancer therapy that have not resolved to Grade ≤1 except for alopecia
* Known, central nervous system (CNS) disease involvement, or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity.
* Evidence of active uncontrolled viral, bacterial, or systemic fungal infection
* Active SARS-CoV-2 infection, irrespective of symptoms.
* History or risk of severe, chronic, untreated, or currently active autoimmune disease
* Prior solid organ transplant or has had an allogenic hematopoietic stem cell transplant within the past 20 years
* Pregnant, lactating, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced an Adverse Event (AE) | 36 months
  An AE is any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. The number of participants who discontinued study treatment due to an AE will be presented.
Number of Dose-Limiting Toxicities (DLTs) | 21 days (cycle 1)
  DLTs will be evaluated according to NCI CTCAE v5.0 and are generally defined as grade 3 or higher toxicities which are deemed to be medically significant.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Profile of Participants Treated with ADA-011 (AUC) | 36 months
  Pharmacokinetic (PK) parameters of ADA-011 including area under the curve (AUC) will be evaluated for all participants in the dose escalation cohorts.
Pharmacokinetic (PK) Profile of Participants Treated with ADA-011 (Cmax) | 36 months
  Pharmacokinetic (PK) parameters of ADA-011 including maximum concentration (Cmax) will be evaluated for all participants in the dose escalation cohorts.

OTHER OUTCOMES:
Number of Participants Positive for Anti-Drug Antibodies (ADA) After Treatment with ADA-011 | 36 months
  Serum samples from participants treated with ADA-011 will be analyzed for ADA using a neutralizing antibody assay. The number of participants with neutralizing ADA will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 36 months
  The percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 criteria will be reported.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - Florida Cancer Specialists, Orlando, Florida
  - Duke University, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon